CLINICAL TRIAL: NCT05012384
Title: Effect of Vergence Exercises for Rehabilitation of Patients With Convergence Insufficiency as a Long-term Consequence of Concussion.
Brief Title: Effect of Vergence Exercises for Patients With Convergence Insufficiency After Concussion.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Danish College of Optometry and Vision Science (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-10-72-22-21
Record Dates: First submitted 2021-07-08; First posted 2021-08-19 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Concussion, Mild; Convergence Insufficiency
MeSH Terms: conditions — Brain Concussion; Ocular Motility Disorders

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vergence exercises (Experimental): Orthoptic vergence exercises
  Interventions: Other: Vergence exercises (Orthoptic exercises)
- Generic treatment (Placebo Comparator)
  Interventions: Genetic: Placebo

INTERVENTIONS:
Other: Vergence exercises (Orthoptic exercises) — Vergence exercises as described by the Convergence Insufficiency Treatment Trials Group (CITT)
  Arms: Vergence exercises
Genetic: Placebo — Generic management plan with non-visual elements
  Arms: Generic treatment

SUMMARY:
A large proportion of concussion patients with long-term consequences of concussion experience visually related symptoms such as headache, blurred vision, double vision, and fatigue.

These patients often have difficulties coordinating the movement of the two eyes (convergence insufficiency) which is essential for single and clear vision to be obtained and is hence a likely explanation for the symptoms.

100 patients with long-term symptoms of concussion and convergence insufficiency will be offered either exercises or placebo treatment the evaluate the effect of exercises aimed at improving coordination between the two eyes.

The study will provide data to support clinicians in deciding whether to use exercises or not as a treatment of symptoms for patients with convergence insufficiency as a long-term consequence of concussion.

ELIGIBILITY:
Inclusion Criteria:

* Concussion at least 3 month ago
* Convergence insufficiency which has not been diagnosed prior to the concussion

Exclusion Criteria:

* Patient who are unable to fulfill baseline examination
* Manifest or paralytic strabismus
* Self-reported eye disease

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Convergence Insufficiency Symptom Survey (CISS) week 18 | Duration (5 minutes) and performed at week 18
  Questionnaire assessing the frequency of eye and visually related symptom during near work
Convergence Insufficiency Symptom Survey (CISS) week 36 | Duration (5 minutes) and performed at week 36
  Questionnaire assessing the frequency of eye and visually related symptom during near work
Near point of convergence - week 18 | Duration (2 minutes) and performed at week 18
  Psychophysical test of the eyes ability to converge
Near point of convergence - week 36 | Duration (2 minutes) and performed at week 36
  Psychophysical test of the eyes ability to converge
Positive fusional vergence at 40 cm - week 18 | Duration (2 minutes) and performed at week 18
  Psychophysical test of the slow fusional adaptation
Positive fusional vergence at 40 cm - week 36 | Duration (2 minutes) and performed at week 36
  Psychophysical test of the slow fusional adaptation
Vergence facility at 40 cm - week 18 | Duration (2 minutes) and performed at week 18
  Psychophysical test of fast fusional adaptation
Vergence facility at 40 cm - week 36 | Duration (2 minutes) and performed at week 36
  Psychophysical test of fast fusional adaptation

SECONDARY OUTCOMES:
Rivermead post-concussional symptoms questionnaire (RPQ) - week 18 | Duration (5 minutes) and performed at week 18
  Questionnaire assessing the frequency of symptoms during activities of daily living
Rivermead post-concussional symptoms questionnaire (RPQ) - week 36 | Duration (5 minutes) and performed at week 36
  Questionnaire assessing the frequency of symptoms during activities of daily living

CONTACTS AND LOCATIONS:
Locations (1):
- Danish College of Optometry and Vision Science, Randers, Central Region, Denmark, Denmark